CLINICAL TRIAL: NCT01952158
Title: Point Prevalence Study of Multidrug-Resistant Organism Carriage by Healthcare Personnel
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 130195; 13-CC-0195
Record Dates: First submitted 2013-09-24; First posted 2013-09-27 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2017-01-13

CONDITIONS: Multidrug Resistance
Keywords: Multidrug-Resistant Organisms; Hospital Infection; Colonization; Healthcare Personnel
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Acquisition and transmission of MDROs in healthcare facilities is a major patient safety problem, afflicting in particular the antibiotic-exposed and immunodeficient patient populations. MDRO-colonized patients require isolation to reduce the risk of transmission to other patients, and frequently develop infections from their colonizing organisms.

Most clinically relevant MDROs are carried in the gastrointestinal tract; thus perirectal cultures are frequently the surveillance method used to screen for these pathogens. Surveillance to identify MDRO colonization allows for anticipation and timely initiation of effective treatment of patients who develop infection.

The precise modes of transmission within hospitals are not known, but contamination of the hands of healthcare personnel, patient care equipment, and the healthcare environment are thought to play major roles in transmitting MDRO. Suboptimal hand hygiene can lead to transmission on the hands of staff to other patients or colonization of their own gastrointestinal tract. Few studies have investigated intestinal colonization of healthcare professionals. Transmission of bacteria by healthcare personnel is thought to occur primarily via contaminated hands; we wonder whether gastrointestinal carriage by healthcare personnel also plays a role in nosocomial spread.

This study will screen a self-referred convenience sample of 400 healthcare personnel who have contact with patients or patient culture specimens for fecal carriage of MDRO at one point in time. A control group of 400 NIH employees or contractors who do not have contact with patients or patient specimens will also be screened. Samples will be linked to questionnaires to assess the exposure of staff members to patients or culture specimens with known MDRO colonization or infection. We will use molecular typing techniques to link healthcare personnel isolates to patient or environmental isolates. Finally, the study will be conducted in such a way as to preserve to the greatest extent possible the anonymity of volunteers, using a system of alphanumeric identifiers and unmanned drop boxes for specimen collection.

DETAILED DESCRIPTION:
Acquisition and transmission of MDROs in healthcare facilities is a major patient safety problem, afflicting in particular the antibiotic-exposed and immunodeficient patient populations. MDRO-colonized patients require isolation to reduce the risk of transmission to other patients, and frequently develop infections from their colonizing organisms.

Most clinically relevant MDROs are carried in the gastrointestinal tract; thus perirectal cultures are frequently the surveillance method used to screen for these pathogens. Surveillance to identify MDRO colonization allows for anticipation and timely initiation of effective treatment of patients who develop infection.

The precise modes of transmission within hospitals are not known, but contamination of the hands of healthcare personnel, patient care equipment, and the healthcare environment are thought to play major roles in transmitting MDRO. Suboptimal hand hygiene can lead to transmission on the hands of staff to other patients or colonization of their own gastrointestinal tract. Few studies have investigated intestinal colonization of healthcare professionals. Transmission of bacteria by healthcare personnel is thought to occur primarily via contaminated hands; we wonder whether gastrointestinal carriage by healthcare personnel also plays a role in nosocomial spread.

This study will screen a self-referred convenience sample of 400 healthcare personnel who have contact with patients or patient culture specimens for fecal carriage of MDRO at one point in time. A control group of 400 NIH employees or contractors who do not have contact with patients or patient specimens will also be screened. Samples will be linked to questionnaires to assess the exposure of staff members to patients or culture specimens with known MDRO colonization or infection. We will use molecular typing techniques to link healthcare personnel isolates to patient or environmental isolates. Finally, the study will be conducted in such a way as to preserve to the greatest extent possible the anonymity of volunteers, using a system of alphanumeric identifiers and unmanned drop boxes for specimen collection.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthcare personnel at the NIH CC who have contact with patients or patient culture specimens will be eligible for study participation. The control group will consist of NIH employees, contractors of the NIH, C or people who work on the Bethesda NIH campus without exposure to patients or patient culture specimens.

EXCLUSION CRITERIA:

Individuals less than 18 years of age and those with any condition that, in the opinion of the principal investigator or designee, contraindicates participation in the study will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2013-09-13; Primary Completion 2013-09-13 (Actual); Study Completion 2017-01-13 (Actual)

PRIMARY OUTCOMES:
Percentage of study participants colonized | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Brooke K Decker, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Munita JM, Arias CA, Murray BE. Enterococcal endocarditis: can we win the war? Curr Infect Dis Rep. 2012 Aug;14(4):339-49. doi: 10.1007/s11908-012-0270-8. PMID 22661339
- [Background] Calfee D, Jenkins SG. Use of active surveillance cultures to detect asymptomatic colonization with carbapenem-resistant Klebsiella pneumoniae in intensive care unit patients. Infect Control Hosp Epidemiol. 2008 Oct;29(10):966-8. doi: 10.1086/590661. PMID 18754738
- [Background] Lane HJ, Blum N, Fee E. Oliver Wendell Holmes (1809-1894) and Ignaz Philipp Semmelweis (1818-1865): preventing the transmission of puerperal fever. Am J Public Health. 2010 Jun;100(6):1008-9. doi: 10.2105/AJPH.2009.185363. Epub 2010 Apr 15. No abstract available. PMID 20395569
- [Derived] Decker BK, Lau AF, Dekker JP, Spalding CD, Sinaii N, Conlan S, Henderson DK, Segre JA, Frank KM, Palmore TN. Healthcare personnel intestinal colonization with multidrug-resistant organisms. Clin Microbiol Infect. 2018 Jan;24(1):82.e1-82.e4. doi: 10.1016/j.cmi.2017.05.010. Epub 2017 May 12. PMID 28506784